CLINICAL TRIAL: NCT05080972
Title: In-the-kNOW (Novel Approaches to Optimizing Women's Health): A Mobile Application to Optimize HIV Prevention and Sexual/Reproductive Health Communication Among Black Women in the Southern U.S.
Brief Title: Mobile HIV Prevention App for Black Women
Acronym: In-the-kNOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Morehouse School of Medicine (Other); Georgia Institute of Technology (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rasheeta Chandler, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002857; 1R34MH128048-01 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-18 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Mobile Phone Use; Hiv; Stigma, Social
MeSH Terms: conditions — Cell Phone Use; Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in-the-kNOW mobile app. (Experimental): Participants will be assigned to the in-the-kNOW mobile app for four (4) months.
  Interventions: Behavioral: in-the-kNOW mobile app
- Control condition. (Active Comparator): Participants will be randomized to receive a one-time virtual women's health counseling session with a healthcare provider.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: in-the-kNOW mobile app — in-the-kNOW is a mobile app with restricted access through a single-use registration code.
  The app will be developed with regular input from Black women enrolled in Atlanta Healthy Start Initiative (AHSI).
  The app will have culturally- and contextually targeted HIV prevention and optimal sexual health messaging.
  Each participant will have 4 months to engage with the app, with e-reminders in time intervals preferred by the participants (a minimum of 3 times per week) via push notifications. During the 4-month study period, participants will receive push notifications to encourage the use of all app domains: My Logger, My Test, My Resources, and My Circle.
  Research staff will complete 2-month check-ins via phone call or video chat with participants.
  Other Names: in-the-kNOW mobile health app
  Arms: in-the-kNOW mobile app.
Behavioral: Control — The control condition will be a one-time virtual women's health counseling session with a healthcare provider. Participants will get information on
  1. Sexual Transmitted Infections (STI)/HIV prevention,
  2. Family planning, and
  3. General health promotion (e.g., exercise and diet).
  The control condition provides access to HIV prevention materials that are publicly available but that do not offer the dynamic and individually customized features of the health communication/new media research approach proposed herein.
  Control group participants will continue to receive the usual care associated with Atlanta Healthy Start Initiative (AHSI) enrollment.
  The control group will not have access to intervention content (e.g. commodity ordering) until after the study has concluded.
  Research staff will complete 2-month check-ins via phone call or video chat with participants.
  Other Names: Regular Care
  Arms: Control condition.

SUMMARY:
Black women have a significantly higher risk of acquiring HIV compared to their non-Black counterparts.

The purpose of this study is to refine and test a mobile HIV Prevention and Reproductive Health app developed specifically for Black women.

DETAILED DESCRIPTION:
The overall goal in implementing this study will be to assess the feasibility, acceptability, and usability of the in-the-kNOW mobile app. The app will be refined using preliminary data obtained through prior research with Black women in which their perspectives towards the use of an HIV and sexual health mobile app were ascertained.

Preliminary data obtained from a Community Advisory Board (CAB), which will consist predominately of Black women will guide refinement of the content and features included within the mobile app, whilst ensuring that the app is tailored towards the needs and perspectives of Black women.

This will be a randomized study with quantitative data collected through surveys, and qualitative data collected through in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* 18-44 years of age
* Self-identify as Black
* Assigned female at birth and identify as female;
* Individuals who qualify for Pre-Exposure Prophylaxis (PrEP) based on the Centers for Disease Control (CDC) criteria (for residence in high HIV incident areas-reside in Fulton, Cobb, Gwinnett, or Dekalb counties)
* Sexually active within the last 6 months
* HIV-negative
* Owner of an Android or IOS smartphone

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Cognitively impaired or Individuals with Impaired Decision-Making Capacity
* Individuals who are not able to clearly understand English

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Assigned female at birth and identify as female
Enrollment: 56 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Retention Rate | 4 months
  Feasibility is assessed with the retention rate of participants in each study arm. Quantitative survey and qualitative interview data to determine acceptability of both the mobile app and the control condition.
Participants' Satisfaction Interview | 4 months
  Acceptability will be assessed through an interview consisting of open-ended questions. There is not a summary score for this qualitative assessment.
  Question sample:
  1. Overall how would you describe your experience using the app
  2. Was the information on the app helpful in providing education on HIV prevention and safe sex?

SECONDARY OUTCOMES:
Participants Completing HIV Testing | 4 months
  Participants will be asked how many times they got a HIV test in the 12-month period before the study and during the 4-month study period. Additionally, research team will quantify home test kit ordering by participants and receive HIV test results from the lab.
Participant's PrEP Intentions and Initiation | 4 months
  Research team will ask participants to indicate whether they initiated PrEP during the 4-month study period on the post-test survey.
Recruiting sources that yielded the largest number of enrolled individuals | 4 months
  Exit interviews and mobile app analytics will determine the Recruiting sources that yielded the largest number of enrolled individuals.
Recruitment methods used for successful enrollment | 4 months
  Exit interviews will determine the successful recruitment methods.
The elapsed time from first contact to enrollment | 4 months
  The research team will use mobile app analytics (e.g., Google Analytics) to assess time elapsed in in-app engagement, from consent time to enrollment.
The amount of app interactions | 4 months
  The research team will use mobile app analytics (e.g., Google Analytics) to assess trends in in-app engagement defined by the number of clicks.
Technological challenges or other connection challenges. | 4 months
  Exit interviews will be audio-recorded and analyzed by the research team
Participants' ownership of smartphones and preferred app formats | 4 months
  Exit interviews will be audio-recorded and analyzed by the research team

CONTACTS AND LOCATIONS:
Overall Officials: Rasheeta Chandler, PhD, RN, Principal Investigator — Nell Hodgson School of Nursing, Emory University
Locations (1):
- Center for Black Women's Wellness, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05080972/ICF_000.pdf